CLINICAL TRIAL: NCT03637634
Title: The Children and Adolescents Nasopharyngeal Carcinoma Survivor Study
Acronym: CANPCSS
Status: Not yet recruiting | Type: Observational
Sponsor: Hai-Qiang Mai,MD,PhD (Other)
Collaborators: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Guangdong Provincial People's Hospital (Other); First Affiliated Hospital of Jinan University (Other); Nanfang Hospital, Southern Medical University (Other); Affiliated Cancer Hospital of Shantou University Medical College (Other); Zhanjiang Cancer Hospital (Unknown); Zhongnan Hospital (Other); First People's Hospital of Foshan (Other); Dongguan People's Hospital (Other Government); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Shenzhen Second People's Hospital (Other); Jiangmen Central Hospital (Other); Yuebei People's Hospital (Other); Hunan Cancer Hospital (Other); Cancer Hospital of Guizhou Province (Other); Fudan University (Other); Fujian Cancer Hospital (Other Government); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The First Affiliated Hospital of Zhengzhou University (Other); Zhejiang Cancer Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); Shandong Cancer Hospital and Institute (Other); Jiangsu Cancer Institute & Hospital (Other); Jiangxi Provincial Cancer Hospital (Other); Second Affiliated Hospital of Nanchang University (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Peking University Cancer Hospital & Institute (Other); Cancer Hospital of Guangxi Medical University (Other); Tongji Hospital (Other)
Responsible Party: Sponsor-Investigator, Hai-Qiang Mai,MD,PhD, Hai-Qiang Mai, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: Childhood NPC
Record Dates: First submitted 2018-08-03; First posted 2018-08-20 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: NPC Patients
Keywords: children and adolescents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood, saliva and tumor specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NPC survivors: Survivors of NPC, diagnosed under 21 years of age, between 1990 and 2030. This project will study children and young adults exposed to specific therapeutic modalities, including radiation, chemotherapy, and/or surgery, for an increased risk of late-occurring events associated with excess mortality and morbidity.
- Sibling Controls: A group of sibling controls will be identified to provide: (1) the ability to make direct comparisons with the survivors, (2) data on outcomes in a non-cancer population, and (3) additional comparison group to determine the consistency of findings between data sources.

SUMMARY:
The Children and Adolescents Nasopharyngeal Carcinoma Survivor Study will investigate the long-term effects of nasopharyngeal carcinoma (NPC) and its associated therapies. A prospective and retrospective cohort study will be conducted through a multi-institutional collaboration. This project will study children and adolescents exposed to specific therapeutic modalities, including radiation, chemotherapy, and/or surgery, who are at increased risk of late-occurring adverse health outcomes. A group of sibling controls will be identified and data collected for comparison purposes.

DETAILED DESCRIPTION:
The study will focus on the following objectives:

* Characterize survivors' health with respect to disease- and treatment-related factors.
* Investigate the consequences of various intensities of exposure to chemotherapy and/or radiation on health outcomes (e.g., cardiovascular, reproductive, second cancers, etc…).
* Compare the mortality experience of survivors with the general population.
* Characterize the health-related behaviors, patterns of medical care, and medical follow-up needs of survivors.
* Describe patterns of familial aggregation of cancer, including known (and variations of) cancer family syndromes.
* Collect and store biologic samples (saliva, blood, second tumor tissue) to correlate with health outcomes and use for future research.

ELIGIBILITY:
Inclusion Criteria:

* Patients or their siblings must be informed of the investigational nature of this study and give written informed consent.

  * Patients with histologically confirmed non-keratinizing nasopharyngeal carcinoma (including differentiated type and undifferentiated type, WHO II or III) before age 21 years at one of participating centers.

Exclusion Criteria:

* Already involved in other blind clinical trial.
* The information of tumour response evaluation and survival data cannot be obtained.

Max Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: NPC patients under 21 years old and their siblings
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) | 5 years
  The OS was defined as the duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up.

SECONDARY OUTCOMES:
Progress-free survival(PFS) | 5 years
  Progress-free survival is calculated from the date of randomization to the date of the first progress at any site or death from any cause or censored at the date of the last follow-up
Locoregional failure-free survival(LRFS) | 5 years
  The LRFS is evaluated and calculated from the date of random assignment until the day of first locoregional relapse or until the date of the last follow-up visit
Distant metastasis-free survival(DMFS) | 5 years
  The DMFS is evaluated and calculated from the date of random assignment until the day of first distant metastases or until the date of the last follow-up visit
Short-term toxic effects assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.0) | 3 months
  The shortterm toxic effects were assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.0)

OTHER OUTCOMES:
Long-term toxicities | Through study completion, an average of half year
  QoL was assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTCQLQ-C30)
Long-term toxicities | Through study completion, an average of half year
  EORTC quality of life questionnaire(QLQ) Head and Neck
Long-term toxicities | Through study completion, an average of half year
  Late Effects Normal Tissue Task Force-Subjective, Objective, Management and Analytic (LENT-SOMA) scoring systems
Growth | Through study completion, an average of half year
  Patients will be monitored for height(in metre)
Growth | Through study completion, an average of half year
  Patients will be monitored for weight(in kilogram)
Growth | Through study completion, an average of half year
  Patients will be monitored for BMI(in kg/m^2)
Sex Development | Through study completion, an average of half year
  secondary sex characteristic survey
Sex Development | Through study completion, an average of half year
  sex hormone(estrogen,testosterone) levels(in nmol/L).
Intelligence Development | Through study completion, an average of half year
  Intelligence quotient by Stanford-Binet test

CONTACTS AND LOCATIONS:
Overall Officials: Hai Mai, Dr, Study Chair — Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center

REFERENCES:
- [Background] Wei WI, Sham JS. Nasopharyngeal carcinoma. Lancet. 2005 Jun 11-17;365(9476):2041-54. doi: 10.1016/S0140-6736(05)66698-6. PMID 15950718
- [Background] Levine PH, Connelly RR, Easton JM. Demographic patterns for nasopharyngeal carcinoma in the United States. Int J Cancer. 1980 Dec 15;26(6):741-8. doi: 10.1002/ijc.2910260607. PMID 7216543
- [Background] Ingersoll L, Woo SY, Donaldson S, Giesler J, Maor MH, Goffinet D, Cangir A, Goepfert H, Oswald MJ, Peters LJ. Nasopharyngeal carcinoma in the young: a combined M.D. Anderson and Stanford experience. Int J Radiat Oncol Biol Phys. 1990 Oct;19(4):881-7. doi: 10.1016/0360-3016(90)90008-8. PMID 2120164
- [Background] Downing NL, Wolden S, Wong P, Petrik DW, Hara W, Le QT. Comparison of treatment results between adult and juvenile nasopharyngeal carcinoma. Int J Radiat Oncol Biol Phys. 2009 Nov 15;75(4):1064-70. doi: 10.1016/j.ijrobp.2008.12.030. Epub 2009 Mar 26. PMID 19327901